CLINICAL TRIAL: NCT04286152
Title: Mirabegron And Ureteral Stent-related Pain (MAP) Trial
Acronym: MAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Urological Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-086
Record Dates: First submitted 2020-02-19; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: This study is a randomized, placebo-controlled, double blinded trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirabegron and narcotic analgesia (Experimental): Drug: Mirabegron 50mg tablet, oral, daily from stent insertion until removal - 7days Drug: Hydromorphone 1mg tablet oral, every 4 hours as necessary Drug: Tylenol ES 500mg tablet , oral, every 6 hours as necessary
  Interventions: Drug: Mirabegron 50 MG
- Placebo (Placebo Comparator): Drug: Placebo for Mirabegron, 1 tablet, oral, daily from stent insertion until removal - 7days Drug:Hydromorphone 1mg tablet oral, every 4 hours as necessary Drug: Tylenol ES 500mg tablet , oral, every 6 hours as necessary
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Mirabegron 50 MG — The experimental drug is administered to patients PO once a day for 7 days from stent insertion until removal
  Other Names: Myrbertiq
  Arms: Mirabegron and narcotic analgesia
Drug: Placebo oral tablet — A sugar pill manufactured to mimic Mirabegron 50 mg tablet is administered to patients PO once a day for 7 days from stent insertion until removal
  Arms: Placebo

SUMMARY:
Ureteric stents are used often following ureteroscopy for prevention of obstruction from edema and/or stone fragments.

Up to 75% of patients experience pain following stenting, as well as lower urinary tract symptoms (LUTS) such as finding blood in the urine, voiding often, the need to urinate quickly resulting in a significant source of morbidity. The negative impact of stents results in a significant impact on health related quality of life.

There is no standard of care for managing ureteric stent pain and lower urinary tract symptoms following surgery. A combination of α-blockers, antimuscarinics, acetaminophen, nonsteroidal anti-inflammatory drugs and opioids are currently the mainstay for treatment of post-operative pain and LUTS following stenting.

Mirabegron is a beta-agonist that mediate relaxation of the detrusor muscle and has been useful in treating overactive bladder (OAB) which has similar symptoms to patients with an ureteric stent in place. Our goal is to assess if mirabegron can improve symptoms and decrease the need for additional pain medications.

The investigators hypothesize that Mirabegron is effective in decreasing ureteral stent related LUTS and pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. First ureteroscopic treatment for the ureteric or renal stone
3. Retrograde semi-rigid or flexible ureteroscopy
4. Placement of a 6Fr, 22-28cm hydrophilic coated ureteric stent
5. Follow-up 7 days post operatively at St. Michael's Hospital
6. Patient who can read and understand English

Exclusion Criteria:

1. Bilateral ureteral stents
2. Stent in situ prior to ureteroscopy
3. Pregnancy or breast feeding, or planning on becoming pregnant in the upcoming weeks
4. Patients with congenital renal abnormalities (eg: pelvic kidney, ureteric duplication) that may impair proper stent placement
5. Patients with urinary diversion or stone in a transplant kidney
6. Patients with a history of interstitial cystitis/painful bladder syndrome, prostatitis, pelvic pain due to other conditions (eg: endometriosis), or neurogenic bladder
7. Indwelling Foley catheter
8. Patients currently taking antimuscarinics, mirabegron, or α-blockers
9. Patients with contraindications to receiving mirabegron (ie: urinary retention, end-stage renal disease, uncontrolled hypertension, known QT prolongation)
10. Significant cognitive impairment
11. Patients with contraindications to opioid use (hypersensitivity, MAO inhibitor use within 14 days, severe respiratory depression, acute or severe asthma, GI obstruction, paralytic ileus, GI stricture)
12. Suspected or confirmed ureteral perforation
13. Stent placement without tether
14. Untreated urinary tract infection
15. Antegrade ureteroscopy
16. Opioid addiction
17. Plan for stent removal at another centre other than St. Michael's Hospital
18. Moderate to severe cardiovascular disease and cerebrovascular disease
19. Signs of hepatic dysfunction including significant liver function test elevation
20. Patients who cannot read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this trial is to assess ureteral stent pain related using a visual analog scale (VAS) and the cumulative score of the 8 pain questions from the Ureteral Stent Symptom Questionnaire (USSQ). | 7 days
  The primary objective of the study is to determine if Mirabegron is effective in decreasing ureteral stent related pain following ureteroscopy when compared to placebo. The visual analog scale (VAS) is a validated, subjective method for measuring pain. The patient makes daily a handwritten mark on a 10-cm line that represents a continuum between 0 ("no pain") and 10 ("worst pain") based on his/her perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point marked by the patient. Pain will also be measured utilizing the "Body Pain" section (questions P1-P9) from the Ureteral Stent Symptoms Questionnaire (USSQ). This is a self-administered questionnaire for patients to report their symptoms for comparison, enabling the comparison between the two treatment arms. Higher scores are associated with greater intensity of symptoms reported.

SECONDARY OUTCOMES:
Opioid consumption | 7 days
  This secondary objective is to determine if Mirabegron is effective in decreasing the opioid consumption in order to tolerate stent pain related. The total opioid consumption will be calculated by counting the number of Hydromorphone tablets used per patient plus the opioid equivalence for the Tylenol ES tablets used.
Quality of life impact of Mirabegron for stent symptoms as measured with the Ureteral Stent Symptoms Questionnaire - USSQ. | 7 days
  This secondary objective is to determine if Mirabegron is effective in improving the urinary symptom score utilizing the Ureteral Stent Symptom Questionnaire - USSQ questions U1-U11 from the USSQ. This is a self-administered questionnaire for patients to report their symptoms for comparison, enabling the comparison between the two treatment arms. Higher scores are associated with greater intensity of symptoms reported. (Time Frame: Measured twice, once at the time of surgery when stent is inserted and secondly at the time the stent is removed occurring 7days later.)
General health score (questions G1-G6 from the Ureteral Stent Symptom Questionnaire - USSQ) | 7 days
  This secondary objective is to determine if Mirabegron is effective in improving the general health score utilizing the Ureteral Stent Symptom Questionnaire - questions G1-G6 from the USSQ. This is a self-administered questionnaire for patients to report their symptoms for comparison, enabling the comparison between the two treatment arms. Higher scores are associated with greater intensity of symptoms reported. (Time Frame: Measured twice, once at the time of surgery when stent is inserted and secondly at the time the stent is removed occurring 7days later.)
Work performance score (questions W1-W7 from the Ureteral Stent Symptom Questionnaire - USSQ) | 7 days
  This secondary objective is to determine if Mirabegron is effective in improving the Work performance score utilizing the Ureteral Stent Symptom Questionnaire - USSQ questions W1-W7 from the USSQ. This is a self-administered questionnaire for patients to report their symptoms for comparison, enabling the comparison between the two treatment arms. Higher scores are associated with greater intensity of symptoms reported. (Time Frame: Measured twice, once at the time of surgery when stent is inserted and secondly at the time the stent is removed occurring 7days later.)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ordon, MD, FRCSC, Principal Investigator — St. Michael's Hospital, Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No